CLINICAL TRIAL: NCT07374978
Title: Effect of Thrombolysis on 30-day Mortality in Intermediate High Risk Pulmonary Patients With Low Bleeding Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD129/2023
Record Dates: First submitted 2025-09-26; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Embolism Subacute Massive; Thrombolytic Therapy
MeSH Terms: interventions — Thrombolytic Therapy; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): This arm will receive standard anticoagulation in the form of intravenous unfractionated heparin
  Interventions: Drug: Unfractionated Heparin IV
- Study group (Active Comparator): This arm will receive thrombolytic therapy in the form of either streptokinase or recombinant tissue plasminogen activator
  Interventions: Drug: Thrombolytic therapy for the study group in the form of streptokinase or recombinant tissue plasminogen activator

INTERVENTIONS:
Drug: Thrombolytic therapy for the study group in the form of streptokinase or recombinant tissue plasminogen activator — Thrombolytic therapy acting on thrombus in pulmonary embolism patients
  Arms: Study group
Drug: Unfractionated Heparin IV — Standard anticoagulation
  Arms: Control group

SUMMARY:
The aim of investigators was to study the effect and safety of Thrombolysis in Intermediate high risk pulmonary embolism patients with low bleeding risk as regards Mortality and bleeding events.

DETAILED DESCRIPTION:
InvestIgators aimed to determine the effect of thrombolysis in Intermediate high risk pulmonary embolism patients with low bleeding risk as regards mortality and bleeding events.

Study design : randomized clinical study conducted Ain Shams University Hospitals over 2 years duration , included 100 participants divided into two groups; control group (50) and study group (50).

Participants assigned to the control group received standard treatment in the form of anticoagulation (intravenous unfractionated heparin) whole participant assigned to control group received thrombolytic therapy (streptokinase or recombinant tissue plasminogen activator) Investigators performed baseline echocardiography for all participants before receiving treatment and assessment of bleeding risk using HASBLED score Follow up of participants' vital data was done in a monitored care unit Participants were assessed one month later for dyspnea and its grade and follow up echocardiography was done also.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermediate high risk pulmonary embolism diagnosed according to clinical probability using revised Geneva Score and diagnosis confirmed by echocardiography and Troponin I or T level and CT pulmonary angiography

Exclusion Criteria:

* o High risk PE

  * Intermediate low risk PE
  * low risk PE
  * Patients with left ventricular systolic dysfunction (ischemic or non-ischemic etiology)
  * Patients with chronic lung diseases (obstructive or restrictive)
  * Patients with contraindications to thrombolysis:
* History of haemorrhagic stroke or stroke of unknown origin
* Ischaemic stroke in previous 6 months
* Central nervous system neoplasm
* Major trauma, surgery, or head injury in previous 3 weeks
* Bleeding diathesis (known inherited bleeding disorder, for example, haemophilia, platelet count <50,000/uL)
* Active bleeding
* Transient ischaemic attack in previous 6 months
* Oral anticoagulation
* Pregnancy or first post-partum week
* Non-compressible puncture sites
* Traumatic resuscitation
* Severe hypertension (systolic BP >180 mmHg)
* Advanced liver disease
* Infective endocarditis
* Active Peptic ulcer
* Patients who develop hypotension or bradycardia or allergic reaction requiring discontinuation of Streptokinase infusion.
* Patients with HAS-BLED score greater than or equals 3 (high bleeding risk for thrombolysis)

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
30 day mortality and bleeding events | 30 days for mortality and bleeding within hospital stay duration
  Cardiac arrest due to pulmonary embolism (mortality) and major bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided